CLINICAL TRIAL: NCT03864510
Title: Evaluating Prevalence and Severity of NAFLD In Primary Care
Brief Title: NAFLD in Diabetes Type 2 in Primary Care
Acronym: EPSONIP
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Mattias Ekstedt, Senior Lecturer/Consultant, Linkoeping University
Other Study IDs: 2018:176-31
Record Dates: First submitted 2019-02-12; First posted 2019-03-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-03

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, RNA, liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The EPSONIP (Evaluating Prevalence and Severity Of NAFLD In Primary care) trial is a longitudinal cohort study of patients with T2DM recruited from primary health care centers in Östergötland, Sweden. The latest MRI techniques will be used to quantify the amount of hepatic fat, inflammation, liver fibrosis and body composition. Each patient will be investigated twice with three years apart to determine patients with progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2
* Age 35-75 year

Exclusion Criteria:

* Contraindication to MR
* Alcohol dependance
* Previously diagnosed liver cirrhosis
* Previously known liver disease (other than fatty liver)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively enrolled patients with diabetes type 2 in primary care.
Sampling Method: Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of fatty liver | 2020
  Number of patients with fatty liver measured with MR-PDFF
Prevalence of advanced liver disease | 2020
  Number of patients with advanced liver disease (fibrosis stage > 2)
The association between physical activity and advanced liver disease (fibrosis >2) | 2020
  Liver fibrosis measured with MRE and liver biopsy. Physical activity measured with the international fitness scale (IFIS)
The association between physical activity and advanced liver disease (fibrosis >2) | 2020
  Liver fibrosis measured with MRE and liver biopsy. Physical activity measured with Actigraph GT3X (accelerometer)
The association between fitness and advanced liver disease (fibrosis >2) | 2020
  Liver fibrosis measured with MRE and liver biopsy. Fitness measured with the six minute walk test.
Genetic factors associated with advanced liver disease (fibrosis >2) | 2020
  Liver fibrosis measured with MRE and liver biopsy. Genes to be analyzed: PNPLA3, TM6SF2, MBOAT

SECONDARY OUTCOMES:
Health economic model for disease management | 2025
  Markow model
Number of patients that develop symptoms of end-stage liver disease | 2030
  Symptoms of end-stage liver disease (ascites, encepahopathy, varices, HCC) or liver related Death will be recorded through chart review

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ekstedt, MD, PhD, Principal Investigator — LiU
Locations (2):
- Sweden (2):
  - Ekholmen primary health care centre, Linköping, Swedish
  - Åby primary health care centre, Norrköping

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bergram M, Kechagias S, Iredahl F, Balkhed W, Holmberg M, Dahlstrom N, Lundberg P, Nasr P, Ekstedt M, Radholm K. Microvascular complications of type 2 diabetes with or without MASLD: the EPSOMIP study, a primary care cohort study. BMC Prim Care. 2025 Nov 11;26(1):354. doi: 10.1186/s12875-025-03096-2. PMID 41219835
- [Derived] Nasr P, Iredahl F, Dahlstrom N, Radholm K, Henriksson P, Cedersund G, Dahlqvist Leinhard O, Ebbers T, Alfredsson J, Carlhall CJ, Lundberg P, Kechagias S, Ekstedt M. Evaluating the prevalence and severity of NAFLD in primary care: the EPSONIP study protocol. BMC Gastroenterol. 2021 Apr 20;21(1):180. doi: 10.1186/s12876-021-01763-z. PMID 33879084